CLINICAL TRIAL: NCT01858753
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled Pilot Study of Azficel-T for the Treatment of Restrictive Burn Scars
Brief Title: Pilot Study of Azficel-T for the Treatment of Restrictive Burn Scars
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unable to enroll
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FI-B-003
Record Dates: First submitted 2013-05-10; First posted 2013-05-21 (Estimated); Results first posted 2021-07-19 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Restrictive Burn Scars
Keywords: burn scars; restrictive; contractures; autologous fibroblasts
MeSH Terms: conditions — Contracture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous fibroblasts (Experimental): Autologous fibroblasts grown in culture from skin biopsy taken from patient. The cells will be injected into the scars to be treated.
  Interventions: Biological: Autologous fibroblasts
- Sterile saline (Placebo Comparator): Sterile saline will be injected into the scar to be evaluated.
  Interventions: Biological: Autologous fibroblasts; Biological: placebo sterile saline

INTERVENTIONS:
Biological: Autologous fibroblasts
  Other Names: Azficel-T
Biological: placebo sterile saline
  Arms: Sterile saline

SUMMARY:
This Phase II, double-blind, randomized, placebo-controlled pilot study is designed to determine whether injection of autologous fibroblasts can increase the mobility (decrease the restriction) of burn scars. The study will assess the effects of azficel-T (autologous fibroblasts) in subjects who have a unilateral burn scar that is no deeper than the fascia (i.e., underlying structures including ligament, tendon, muscle, and bone must not contribute to the restriction) and that is either:

1. An axillary scar causing 20-60% restriction of shoulder adduction
2. An anterior elbow scar causing 20-60% restriction of elbow extension
3. A dorsal or palmar lesion of a single finger causing 20-60% restriction of flexion or extension

Subjects will each receive 2 injections of azficel-T or placebo administered 14 days (± 7 days) apart (depending on cell availability) and will be followed for efficacy (including range of motion measurements, scar pain and ability to perform activities) to Visit 7 and for safety to Visit 9 at 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject has a unilateral burn scar of a jointed area (i.e., finger, elbow, shoulder) that is no deeper than the fascia (i.e., underlying structures including ligament, tendon, muscle, and bone must not contribute to the restriction) and that is either:

   1. An axillary scar causing 20-60% restriction of shoulder abduction
   2. An anterior elbow scar causing 20-60% restriction of elbow extension
   3. A dorsal or palmar lesion of a single finger causing 20-60% restriction of flexion or extension
3. Subject's burn scar to be treated is <100 sq cm in size
4. Injury occurred ≤ 36 months prior to screening
5. By the Investigator's assessment, physical therapy will not provide significant continuous improvement to the range of motion of the subject's joint
6. Subject agrees to maintain any current physical therapy regimen for the duration of the study
7. Subject must be able to provide written informed consent and comply with the study requirements
8. Females of childbearing potential must have a negative urine pregnancy test at the screening visit and prior to the first treatment, and must agree to use a reliable means of birth control for the duration of the study
9. Subject has healthy, non-scarred post auricular skin area suitable for biopsy
10. Subject must have a normal complete blood count (CBC) and chemistry panel within 90 days prior to enrollment

Exclusion Criteria:

1. Restrictive burn scars that are primarily classified as keloid scars
2. Subjects for whom a post auricular biopsy cannot be collected for azficel-T production
3. Sunburn or sun damage in the area that will be used for biopsy
4. Plans to initiate any other new scar therapy during the study period
5. Treatment with an investigational product or procedure within 30 days prior to study enrollment or plans to participate in another clinical trial during the course of this study
6. History of active autoimmune disease or organ transplantation
7. Diagnosis of cancer, including basal cell carcinoma, unless successfully treated or in remission for a minimum of 6 months
8. Known genetic disorders affecting fibroblasts or collagen, such as achondroplasia, osteogenesis imperfecta, epidermolysis bullosa, ataxia-telangiectasia, Ehlers Danlos syndrome, etc.
9. Active systemic infection
10. Requires chronic antibiotic or steroidal therapy
11. Any conditions that are considered by the Investigator to be contraindications to biopsy or injection
12. Pregnant or lactating women, or women trying to become pregnant during the study
13. Subject has any disorder that may prevent compliance, such as history of chronic alcohol or drug abuse, significant mental or nervous disorder or other illness that would, in the Investigator's opinion, interfere with the study
14. Presence of other disease or condition that would result in impairment of the range of motion of the extremity, e.g., rheumatoid arthritis or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Lozano, MD, Principal Investigator — Lehigh Valley Health Network
Locations (9):
- United States (9):
  - Univ of California David Medical Center, Sacramento, California
  - Univ of California San Diego, San Diego, California
  - Division of Burns and Trauma, Jackson Memorial Hospital, Miami, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Richard M. Fairbanks Burn Center, Indianapolis, Indiana
  - Long Island Plastic Surgical Group, Garden City, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Center for Innovation in Restorative Medicine, Pittsburgh, Pennsylvania
  - Univ of Washington, Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were screened to determine eligibility for the study prior to enrollment. Once the subjects were enrolled, the biopsy was performed within 14 days after screening. Subjects were then randomized sequentially as their cells were harvested and found to be acceptable.
Groups:
- Autologous Fibroblasts: Autologous fibroblasts grown in culture from skin biopsy taken from patient. The cells will be injected into the scars to be treated.
  Autologous fibroblasts
- Sterile Saline: Sterile saline will be injected into the scar to be evaluated.
  Autologous fibroblasts
  placebo sterile saline
Period: Overall Study
Arm/Group | Autologous Fibroblasts | Sterile Saline
Started | 5 | 0
Completed | 0 | 0
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Population: MITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Fibroblasts | Sterile Saline | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (13.00) |  | 56.0 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 3 |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3
ROM of the Affected Joint [Mean (Standard Deviation); unit: degrees] | 124.0 (39.34) |  | 124.0 (39.34)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline (CFB) of Range of Motion (ROM) of the Affected Joint
Description: Percentage CFB was calculated by subtracting the baseline ROM measurement from the post-treatment ROM measurement, divided by the baseline ROM measurement, and multiplying by 100.
Time Frame: Baseline and post-treatment (visit occurred between 194 - 208 days from baseline)
Population: Modified intent to treat population (mITT)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Autologous Fibroblasts | Sterile Saline
Number analyzed (Participants) | 3 | 0
percent change | 52.0 (23.40) |

2. Primary Outcome: Percentage CFB of ROM of the Affected Joint
Description: as for outcome 1
Time Frame: Baseline and post-treatment (visit occurred between 23 - 37 days from baseline)
Population: Modified intent to treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Autologous Fibroblasts | Sterile Saline
Number analyzed (Participants) | 3 | 0
percent change | 39.6 (10.88) |

3. Primary Outcome: Percentage CFB of ROM of the Affected Joint
Description: as for outcome 1
Time Frame: Baseline and post-treatment (visit occurred between 53 - 67 days from baseline)
Population: Modified intent to treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Autologous Fibroblasts | Sterile Saline
Number analyzed (Participants) | 3 | 0
percent change | 54.9 (25.86) |

4. Primary Outcome: Percentage CFB of ROM of the Affected Joint
Description: as for outcome 1
Time Frame: Baseline and post-treatment (visit occurred between 93 - 97 days from baseline)
Population: Modified intent to treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Autologous Fibroblasts | Sterile Saline
Number analyzed (Participants) | 3 | 0
percent change | 56.0 (29.33) |

5. Primary Outcome: Percentage CFB of ROM of the Affected Joint
Description: as for outcome 1
Time Frame: Baseline and post-treatment (visit occurred between 113 - 127 days from baseline)
Population: Modified intent to treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Autologous Fibroblasts | Sterile Saline
Number analyzed (Participants) | 3 | 0
percent change | 52.0 (23.40) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of the subject's biopsy through visit 9 (i.e., 360 days from their second treatment).
Arm/Group | Autologous Fibroblasts | Sterile Saline
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 2/5 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Autologous Fibroblasts (N=5) | Sterile Saline (N=0)
Injection site pain (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects enrolled and completed; some data uninterpretable due to late data entry. With low enrollment (three subjects in mITT population and five subjects in safety population), a meaningful statistical analysis was not possible for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No